CLINICAL TRIAL: NCT00801463
Title: Prednisone Plus Tripterygium Wilfordii Treatment of Adult Patients With Idiopathic Focal Segmental Glomerulosclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine, Research Institute of Nephrology, Jinling Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NJCT-0801
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2009-04

CONDITIONS: Proteinuria; Focal Segmental Glomerulosclerosis
Keywords: Focal Segmental Glomerulosclerosis; Prednisone; Tripterygium Wilfordii
MeSH Terms: conditions — Proteinuria; Glomerulosclerosis, Focal Segmental

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Large pred (Experimental): Prednisone 60mg/d*8 wks
  Interventions: Drug: tripterygium wilfordii (TW)
- small pred (Experimental): Pred 30mg/d*8wks
  Interventions: Drug: tripterygium wilfordii (TW)

INTERVENTIONS:
Drug: tripterygium wilfordii (TW) — Pre 30mg/d +TW 120 mg/d, po for 12 weeks
  Other Names: tripterygium wilfordii

SUMMARY:
The purpose of this study is to assess the efficacy of prednisone and tripterygium wilfordii in treated Focal Segmental Glomerulosclerosis (FSGS).

DETAILED DESCRIPTION:
Primary FSGS is a leading cause of end stage renal disease in adults, with complete loss of kidney function in 50% of patients over 10 years. Steroids, which are currently used to treat the disease, are effective in part of patients. Over the past decade, a number of studies have reported therapeutic efficacy for treatment with high-dose and over 6mo prednisone in patients with FSGS. These studies show that the total effective rates were only around 50%. But this therapy had taken some side effects of prednisone. Except these studies, in recent studies suggest that Tripterygium Wilfordii may be effective for passive Heymann nephritis, podocyte injury in nephrosis rats induced y puromycin aminonucleoside, and so on. FSGS is a podocytepathy. There was no-data of Prednisone and Tripterygium Wilfordii treatment of Chinese adult patients with idiopathic FSGS.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years at onset of signs or symptoms of FSGS
* Urine protein ≥ 3.5 g/24 h
* Estimated glomerular filtration rate (GFR) ≥ 40 ml/min/1.73 m2, serum creatinine<2.5mg/dl
* Biopsy confirmed as idiopathic FSGS (including all subtypes)
* Willingness to follow the clinical trial protocol, including medications, and baseline and follow-up visits and procedures

Exclusion Criteria:

* Secondary FSGS
* Prior therapy with sirolimus, Cyclosporine, MMF, azathioprin, cytoxan, chlorambucil, levamisole, methotrexate, or nitrogen mustard in the last 90 days
* Active/serious infection
* Malignancy
* Previously diagnosed as diabetes mellitus type 1 or 2, or abnormal carbohydrate tolerance
* Peripheral white blood cells < 3000/ul
* Clinical evidence of cirrhosis or chronic active liver diseases
* History of significant gastrointestinal disorder
* Allergy to study medications, and Inability to consent/assent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2009-01; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy and safety of TW in the treatment of FSGS | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-hong Liu, M.D, Principal Investigator — Research Institute of Nephrology, Jinling Hospital,
Locations (1):
- Research Institute of Nephrology, Jinling Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Hodson EM, Sinha A, Cooper TE. Interventions for focal segmental glomerulosclerosis in adults. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD003233. doi: 10.1002/14651858.CD003233.pub3. PMID 35224732